CLINICAL TRIAL: NCT06951958
Title: The Effect of Cardiac Rehabilitation Program Based on Health Action Process Approach Model on Treatment Compliance, Quality of Life and Functional Capacity Level in Individuals With Myocardial Infarction
Brief Title: Application of the Health Action Process Approach Model Program to Patients With Heart Attacks
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gönül Taşcı, PhD student, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GTasci
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Heart Attack Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Behavioral Interventions will be provided to the intervention group using the Cardiac Rehabilitation Program based on the Health Action Process Approach Model.
  Interventions: Behavioral: Cardiac Rehabilitation Program Based on Health Action Process Approach Model
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation Program Based on Health Action Process Approach Model — The intervention program will start in the hospital setting and continue at home. A work schedule will be created with each individual in intervention group 1 by determining the times when they are available separately. Individuals are planned to receive 60-minute home visits once a week. In the following weeks, care interventions such as home visits, training, counseling and monitoring will be organized according to the specific needs and requirements of each individual. In the face-to-face preparation phase, the patient's health needs will be identified, health status will be assessed, daily activities will be reviewed, incompatibility between activity levels and recommended exercise guidelines will be examined, and individualized exercise goals and a behavior-specific exercise program will be created for behavioral changes. In the intervention phase, the parts that the patient lacks will be determined and the trainings needed will be given.
  Arms: Intervention group

SUMMARY:
This research is conducted to determine whether the nurse-led Health Action Process Approach Model-based Cardiac Rehabilitation Program is effective in patients with myocardial infarction. The population of the study will consist of coronary angiography patients with myocardial infarction in the cardiology service of a state hospital. In this study, which is planned as a randomized controlled experimental model, 35 intervention and 35 control groups will be studied. As data collection tools; patient identification form, Laboratory Investigations Monitoring Form, Perceived Stress Scale, Health Action Process Approach Based Participant Assessment Form, Health Action Process Approach Based Myocardial Infarction Risk Factors Participant Assessment Form Functional Capacity Assessment Form, Myocardial Infarction Dimensional Assessment Scale and Turkish Modified Morisky Scale will be used. Health Action Process Approach Modeled Cardiac Rehabilitation Program will be applied to the intervention group and no intervention will be applied to the control group. Data will be collected with data collection tools at 6, 12, 24 weeks. SPSS 25.0 (Stastical Package for Social Science) package program will be used for statistical analysis of the data. Descriptive statistics will be given as number, percentage, mean, standard deviation and median values. The normal distribution of the data of numerical variables will be evaluated by Shapiro Wilk test. Two group comparisons will be made with independent two sample t-test for normally distributed variables and with Mann-Whitney U test for variables that do not show normal distribution. Comparisons of the groups' pre-test, week 6, week 18 and week 24 scale scores will be made with two-way analysis of variance in repeated measures from general linear models.

ELIGIBILITY:
Inclusion Criteria:

* To be between 18-70 years old,
* Becoming literate,
* Living in the city center
* Having had a heart attack within the last month,
* Not having had a heart attack before,
* Dyspnea less than 4-5 degrees according to the modified Borg Scale
* No deformity or diagnosis related to the musculoskeletal system that may prevent physical activity, no orthopedic limitation
* Stable New York Heart Association (NHYA) functional class I or II coronary artery disease with myocardial infarction

Exclusion Criteria:

Those with communication disabilities such as speech, vision, hearing

* Dyspnea score of more than 4-5 degrees according to the modified Borg Scale
* Those who stayed in intensive care for a long time after MI
* Complications related to treatment and interventions after MI
* Those who underwent surgical treatment after MI,
* Those with chronic diseases (chronic obstructive pulmonary disease, chronic renal failure, hypertension, diabetes, pulmonary emphysema, rheumatic valve disease, cancer diagnosis, etc.)
* Those who indicated that they would not participate in intervention programs due to time constraints.
* Failure of the six-minute walk test

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Changes in treatment compliance of people participating in the Health Action Process Approach Model-based Cardiac Rehabilitation Program | At the beginning of the study (week 0), week 6, week 12 and week 24
  It was developed by Morisky et al. in 1986. It is a 6-item scale used to measure medication compliance in patients.

SECONDARY OUTCOMES:
Changes in the Quality of Life of People Participating in a Cardiac Rehabilitation Program Based on the Health Action Process Approach Model | At the beginning of the study (week 0), week 6, week 12 and week 24
  Developed in 2002 by Thompson et al, this scale is specific for patients with myocardial infarction. It is a 35-item scale used to measure quality of life in patients.

IPD SHARING:
Plan to Share IPD: No